CLINICAL TRIAL: NCT01521208
Title: LUcas Continuous Chest Compressions in Out-of-hospital Cardiac Arrest Treatment. The LUCAT Trial
Brief Title: LUCAS Chest Compressor Versus Manual Chest Compression in Out-of-hospital Sudden Cardiac Arrest. LUCAT Trial
Acronym: LUCAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sistema d'Emergències Mèdiques (Other Government)
Collaborators: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Francesc Carmona Jimenez, Assistant Investigator, Sistema d'Emergències Mèdiques
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEM-HVH-001
Record Dates: First submitted 2011-12-25; First posted 2012-01-30 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Sudden Cardiac Arrest
Keywords: Out-of-Hospital cardiac arrest (OHCA); Chest compressions; LUCAS device
MeSH Terms: conditions — Death, Sudden, Cardiac; Out-of-Hospital Cardiac Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LUCAS, Continuous chest compressions (Active Comparator): Mechanical continuous chest compressions performed by LUCAS device (also during defibrillation)
  Interventions: Device: LUCAS (Lund University Cardiac Assist Sysrem)
- Manual chest compressions (Active Comparator): Manual chest compression is performed, chest compressions halted during defibrillation
  Interventions: Other: Manual chest compressions

INTERVENTIONS:
Device: LUCAS (Lund University Cardiac Assist Sysrem) — LUCAS device will be placed on patients suffering a cardiac arrest and continuous chest compressions will be performed, even while defibrillation is being applied
  Other Names: Mechanical continuous chest compressions
  Arms: LUCAS, Continuous chest compressions
Other: Manual chest compressions — Manual CPR according to 2010 ERC guidelines will be performed
  Other Names: Cardiopulmonary resuscitation
  Arms: Manual chest compressions

SUMMARY:
The goal of this study is to show the superiority in survival at hospital admittance and in neurological outcome on hospital discharge of continuous mechanical chest compression using LUCAS device versus manual chest compressions in patients who suffered an out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
The primary goals of the trial are:

* To show a survival increase at hospital admittance after out-of-hospital cardiac arrest of patients treated by continuous chest compressions LUCAS device compared with patients treated by manual chest compressions.
* To evaluate neurological outcome on hospital discharge, in two centres (Vall d'Hebron Hospital and Josep Trueta Hospital).

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 80 years ,
* Suffering from NON traumatic or an unexpected SCA,
* SCA witnessed (seen, heard or monitored),
* Attended by an advanced support ambulance (served by doctor or nurse) in Barcelona city, or in the Girona or Lleida area
* Time between alarm-call to SEM 061 and reaching patient is less than 12 minutes.

Exclusion Criteria:

* Biological signs of death
* Age under 18 or over 80 years
* Trauma caused cardio respiratory arrest (CRA), including hanging
* Secondary CRA or intoxication
* Return of spontaneous circulation previous to arrival of SEM's medical team
* Known pregnancy
* Inadequate size for LUCAS device
* Anything in the study that can delay treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Survival at hospital admittance | 2 hours
  The primary goal is to evaluate survival at hospital admittance of patients, after out-of hospital cardiac arrest treated by LUCAS device chest compressions, compared with those patients treated by manual chest compressions
Survival on discharge from hospital (or 30 days if not applicable) in acceptable neurological state (CPC scale 1 or 2) | 30 days
  Evaluate the neurological outcome on hospital discharge, in two centres (Vall d'Hebron Hospital in Barcelona and Josep Trueta Hospital in Girona) 1 or 2 in Cerebral Performance Category

SECONDARY OUTCOMES:
Restoration of spontaneous circulation | 2 hours
  To compare the return of spontaneous circulation (ROSC) between both groups
EndTidal CO2 values | Every four minutes during resuscitation maneuvers
  To compare EndTidal CO2 values of patients during cardiopulmonary resuscitation (CPR)between boths study arms
SOFA scale values | During the first three days and on hospital discharge
  To compare the first three days, on hospital discharge SOFA scale value and the worse value obtained (date and hour) in patients who survived out-of-hospital SCA and weere brought to either Vall d'Hebron Hospital or Josep Trueta Hospital.
Days before discharge from Intensive Care Unit (ICU) / Coronary Care Unit (CCU) | 30 days
  To compare days before discharge from Intensive Care Unit (ICU) / Coronary Care Unit (CCU) in patients who survived out-of-hospital SCA and were brought to either Vall d'Hebron Hospital or Josep Trueta Hospital
Metabolic (pH, lactate) and inflamatory (leukocytes, C reactive protein) parameters | During the first 24h, at >48h and at 5-7days
  To establish the differences in metabolic (pH, lactate) and inflamatory (leukocytes, C reactive protein) parameters in patients who survived out-of-hospital SCA and were brought to either Vall d'Hebron Hospital or Josep Trueta Hospital
Epidemiology of Out-of-Hospital Cardiac Arrest | 3 months
  To describe the epidemiology of out-of-hospital SCA in the cities of Barcelona, Girona and Lleida
To obtain a blood sample for genetic and biological studies | 7 days
  Blood samples from SCA survivors will be kept to perform biological studies.
Left ventricular function | During the first 24h and during the 24h previous on hospital discharge or at two months
  To compare left ventricular function in patients who survived at out-of-hospital sudden cardiac arrest and were brought to either Vall d'Hebron Hospital or Josep Trueta Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Palma Padró, Doctor, Study Director — Sistema d'Emergències Mèdiques
Locations (2):
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - Sistema d'Emergències Mèdiques, L'Hospitalet de Llobregat, Barcelona